CLINICAL TRIAL: NCT03828825
Title: Prospective Evaluation of the Efficacy and Safety of a Simplified Procedure for the Percutaneous Closure of the Patent Foramen Ovale
Brief Title: Evaluation of the Efficacy and Safety of a Simplified Procedure for the Percutaneous Closure of the Patent Foramen Ovale
Acronym: IDFFOP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDFFOP
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Patent Foramen Ovale
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patent Foramen Ovale Closure (Experimental): The percutaneous closure of Patent Foramen Ovale is realized under trans-thoracic echocardiography control. If necessary, the operator will use trans-esophageal echocardiography to implant the prosthesis.
  Interventions: Other: Patent Foramen Ovale closure

INTERVENTIONS:
Other: Patent Foramen Ovale closure — The Patent Foramen Ovale closure is realized under trans-thoracic echocardiography control. If necessary, the operator will use trans-esophageal echocardiography to implant the prosthesis. One day after the procedure, a clinical assessment and an electrocardiogram are performed. At 3 months the consultation corresponds to a trans-thoracic echocardiography validation of the closure accompanied by a "bubble test" (Valsalva maneuver) and a clinical assessment. At 12 months, the visit corresponds to a consultation with a clinical assessment and an electrocardiogram. At 36-months and 60-months, the visits will be done following the on-site visits provided for in the usual care or during a telephone call from the attending cardiologist to retrieve the results of the clinical examination, electrocardiogram and MACCE (major cardiac and cerebral vascular events). A consultation dedicated to the study may be proposed to patients according to what is provided in the usual care.

SUMMARY:
Patent Foramen Ovale, is an embryonic remnant, formed by apposition of the septum primum and septum secondum composing the interatrial septum. This foramen ovale is permeable during intra-uterine life and allows inter-auricular communication. It tends to close at birth, due to increased pressure from the left atrium. However, it remains permeable in almost 25% of the general population. Several studies have shown that this cardiac "anomaly" associated with the atrial septum aneurysm (ASA), easily diagnosed by ultrasound, is more common in patients with cryptogenic stroke. The diagnosis of patent foramen ovale is performed by a cardiac ultrasound with a "bubble" test: a volume of micro-bubbles obtained by emulsion of saline (9 ml) and air (1 ml) is injected intravenously. The path of these microbubbles is observed by trans-thoracic ultrasound and can detect a shunt right / left. This test can be sensitized by Valsalva maneuver and / or cough. The shunt is quantified by the number of microbubbles flowing through the right / left shunt: positive diagnosis: more than 3 bubbles passing; minimal shunt <10 bubbles, moderate shunt between 10 and 30 bubbles, massive shunt if> 30 bubbles.

Patent Foramen Ovale Closure is an interventional cardiac catheterization procedure by venous femoral approach. Several clinical trials show that Patent Foramen Ovale closure prevents stroke recurrence in young people and that this procedure is more effective than antiplatelet therapy. Nevertheless, an increase in the incidence of peri-procedural atrial fibrillation has been observed. For some researchers, this would be explained by irritation of the atrial muscle due to the establishment of the device.

To date, only percutaneous closures made in clinical trials have been evaluated. In fact, there are no specific recommendations. The use in clinical practice of this percutaneous treatment therefore requires an evaluation of the indications but also the profile of the patients to optimize these procedures and reduce the complication rate.

The closure technique and the choice of the size of the prosthesis are not standardized. The closure is done under trans-esophageal echocardiography (invasive method) or trans-thoracic echocardiography (non-invasive method) depending on the choice of the practitioner. In CLOSE study, this rate is not specified. The procedure rate under general anesthesia is 54%. This category of patients can be assumed to use a trans-esophageal echocardiography.

The absence of specific recommendations concerning the technical modalities of this procedure lead us to study the closure of Patent Foramen Ovale standardized under trans-thoracic echocardiography and to evaluate its possible reliefs by avoiding the general anesthesia and the use of trans-esophageal echocardiography. The objective of the study is to bring elements of standardization of the technique. As part of a "real life" study, we will evaluate the success rate of procedure under local anesthesia and under trans-thoracic echocardiography control. This evaluation will be done by trans-thoracic echocardiography at 3 months, the re-endothelisation time of the medical device being between 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient with cryptogenic ischemic stroke
* Patient with FOP / ASA in trans-esophageal echocardiography
* Patient with spontaneous and / or induced Shunt R/L
* ROPE score> 5
* Patient with medical insurance
* Francophone patient
* Patient giving free, informed and express consent

Exclusion Criteria:

* Patient with a stroke with known etiology
* Patient with atrial fibrillation
* Patient with emboligenic heart disease
* Patient with carotid stenosis
* Patient with infectious endocarditis
* Patient with uncontrolled hypertension
* Patient for whom the percutaneous closure of the FOP is performed by a medical device under evaluation
* Patient under tutorship or curatorship
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of a simplified procedure for the percutaneous closure of the Patent Foramen Ovale | Month 3
  Rate of disappearance of shunt Right / Left (D / G) by trans-thoracic echocardiography control

SECONDARY OUTCOMES:
Safety of a simplified procedure for the percutaneous closure of the Patent Foramen Ovale | during the procedure
  Rate of peri-procedural complications
Safety of a simplified procedure for the percutaneous closure of the Patent Foramen Ovale at 1 month | Month 1
  Rate of complications
Safety of a simplified procedure for the percutaneous closure of the Patent Foramen Ovale | Year 1
  Rate of complications
Safety of a simplified procedure for the percutaneous closure of the Patent Foramen Ovale | Year 3
  Rate of complications MACCE
Safety of a simplified procedure for the percutaneous closure of the Patent Foramen Ovale | Year 5
  Rate of complications MACCE
Evaluation of the frequency of cases where a procedural "switch" | during procedure
  Patients number for whom procedural "switch" (trans-thoracic echocardiography control discontinuation with trans-esophageal echocardiography) will be required

CONTACTS AND LOCATIONS:
Overall Officials: Pryscille KAMTCHUENG, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (3):
- France (3):
  - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - Centre Cardiologique du Nord, Saint-Denis